CLINICAL TRIAL: NCT06854744
Title: Zinc Oxide Ozonated Oil Versus Modified Triple Antibiotic Paste as a Lesion Sterilization and Tissue Repair Technique in Primary Molars
Brief Title: Zinc Oxide Ozonated Olive Oil in LSTR
Acronym: Zn-OO/MTAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nouran Esmail Mohamed Shalaby, Zinc Oxide Ozonated Oil Versus Modified Triple Antibiotic Paste as a Lesion Sterilization and Tissue Repair Technique in Primary Molars, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-23-2093
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Irreversible; Ozone; Pulp Disease, Dental; Primary Teeth
Keywords: ZnOO /MTAP
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Wound Healing

STUDY DESIGN:
Intervention Model Description: This study will be carried out to evaluate and compare the clinical and radiographic effect of zinc oxide-ozonated olive oil (ZnO-OO) versus Modified Triple Antibiotic Paste (MTAP) as a Lesion Sterilization and Tissue Repair Technique in Primary Molars
Who Masked: Participant
Masking Description: Group I: Zinc Oxide Ozonated Olive- oil will be applied to the pulp stamps of the molars on one side.
  Group II: MTAP will be applied to the pulp stamps of the molars on the other side.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc Oxide Ozonated Oil (Experimental): Zinc Oxide Ozonated Oil as a Lesion Sterilization and Tissue Repair Technique in Primary Molars
  Interventions: Procedure: lesion sterlization and tissue repair; Other: Zinc Oxide Ozonated Oil
- Modified Triple Antibiotic Paste (Experimental): Modified Triple Antibiotic Paste (MTAP)as a Lesion Sterilization and Tissue Repair Technique in Primary Molars
  Interventions: Procedure: lesion sterlization and tissue repair; Other: Modified Triple Antibiotic Paste

INTERVENTIONS:
Procedure: lesion sterlization and tissue repair — evaluate and compare the clinical and radiographic effect of zinc oxide-ozonated olive oil (ZnO-OO) versus Modified Triple Antibiotic Paste (MTAP) as a Lesion Sterilization and Tissue Repair Technique in Primary Molars.
  Other Names: zinc oxide ozonated oil and modified triple antibiotic paste
Other: Zinc Oxide Ozonated Oil — Zinc Oxide Ozonated Oil
  Arms: Zinc Oxide Ozonated Oil
Other: Modified Triple Antibiotic Paste — Modified Triple Antibiotic Paste
  Arms: Modified Triple Antibiotic Paste

SUMMARY:
This study will be carried out to evaluate and compare the clinical and radiographic effect of zinc oxide-ozonated olive oil (ZnO-OO) versus Modified Triple Antibiotic Paste (MTAP) as a Lesion Sterilization and Tissue Repair Technique in Primary Molars

DETAILED DESCRIPTION:
Preservation of primary dentition is crucial for the development of arch form, esthetics, function, mastication, and normal eruption of permanent teeth. Premature loss, especially of the primary second molar, can cause several problems. The first permanent molars typically erupt mesially as a result, leading to some problems including the ectopic eruption of the second premolar, the loss of space for the succeeding permanent teeth and functional impairment 1.

Dental caries is the most prevalent non-communicable disease in children with significant aesthetic, functional, and quality of life deterioration2. Caries lesions can jeopardize the teeth' vitality, as their progression cause infection, pain, and even early tooth loss 2,3. Thus, timely intervention is key to avoid unfavorable repercussions for the child. Depending on the depth of caries (which may have pulp involvement), two approaches may be considered in the primary dentition: vital pulp therapy (VPT) or non-vital therapy (NPT)2,4.

When the pulp can be recovered, VPT may be an option and three options are available: indirect pulp treatment (IPT), direct pulp cap (DPC), and pulpotomy 2-6.

When the caries lesion progresses to the point where the pulp necrotizes, then an NPT is performed, such as a pulpectomy 4. It is a nonvital treatment (NVT), a root canal treatment with irreversibly inflamed or necrotic pulp resulting from caries or trauma 2,4,6,7. Pulpectomy has been the gold-standard treatment for primary teeth with pulp necrosis or irreversible pulp inflammation and is based on the debridement of the root canals with manual or rotary instruments together with the use of antimicrobial irrigation solutions to decontaminate the root canal system for posterior filling with resorbable materials 8 However, the inherent characteristics of the root canal system in primary teeth make this procedure an endodontic challenge, especially in molars 9,10.

In the 1990s, an innovative procedure called lesion sterilization and tissue repair (LSTR) was proposed as an alternative biologic approach that was thought to facilitate the disinfection of dentinal carious lesions, pulp, and periapical lesions in primary teeth 11-13 with the advantages of being simpler and faster 14,15.

The LSTR is a minimally invasive endodontic therapy method that involves the introduction of an antibiotic combination in a propylene glycol vehicle to disinfect root canal systems and periapical lesions 16. It is also known as no instrumental endodontic treatment (NIET) 17. The rationale of LSTR is that combination of three antibiotics (3Mix) can sterilize necrotic pulps and infected root dentine of primary teeth. In primary dentition, LSTR has shown a high rate of clinical success as a substitute for pulpectomy 14,18.

A single antibiotic is insufficient to eradicate pathogenic flora; hence a combination of drugs popularly known as ''triple antibiotic paste'' (TAP) is recommended. This mix is potently active against a wide range of bacteria. It aids in disinfecting and sterilizing the root canal system. It also allows the entry and growth of new tissue in the radicular area in regenerative therapy in the case of young, immature teeth. TAP can also assist in the development of a discipline that will allow for the successful application of other desired and necessary therapies 19,20.

Most commonly, a combination of three broad-spectrum antibiotics, namely, ciprofloxacin, metronidazole and minocycline are used for root canal disinfection. Metronidazole acts against obligate anaerobes, which are the most commonly isolated species from infected root canals. Minocycline is a bacteriostatic long-acting antibiotic, potent against a wide range of microorganisms. Ciprofloxacin is added to eradicate Gram-negative species21,22.

The use of cefaclor (a second-generation cephalosporin) instead of minocycline and ornidazole instead of metronidazole in 3Mix improves clinical outcomes 23,24.

Cruz et al. 25 showed that the incorporation of propylene glycol and macrogol (MP) as a carrier vehicle dramatically raised the penetration of these drugs.

Herbal and natural extracts employed in dentistry as irrigants and intracanal medicaments have gained popularity in recent decades because of their antimicrobial activity, biocompatibility, and anti-inflammatory and anti-oxidant properties 26.

New generations of disinfecting agents have been developed among them is ozone, which is a powerful oxidizing agent and can be used to eliminate bacteria in root canals 27.

Ozone's antibacterial impact gets triggered by oxygenated radicals in aqueous solutions, this will cause changes in the osmotic permeability of the cell membranes resulting in cell damage 28. Ozone is not only an antimicrobial agent, but it can also enhance blood circulation and immune response. It can modulate the cellular and humoral immune system of the patient by the proliferation of immunocompetent cells and the synthesis of immunoglobulins. It can stimulate the phagocytosis process, activate the macrophages, and increase the sensitivity of microorganisms to macrophages29.

There are multiple forms for the application of ozone as ozone gas, ozonated water, and ozonated oil that are used for root canal irrigation and as intra-canal medicaments to obtain disinfection of root canal systems. Ozonated water and olive oil act by entrapping ozone and then emitting it 30.

Nowadays, ozone is utilized in the manufacturing of ozonated olive oil (Oleozon), which is increasingly being utilized as a clinical therapeutic agent for wound healing 31.

Olive oil has anti-inflammatory and antibacterial properties, mainly due to its fatty acid's oleic acid and linoleic acid, and its polyphenol compounds, such as hydroxytyrosol, tyrosol, oleuropein, and oleocanthal 32.

Up to our knowledge, no previous studies discussed Zinc oxide-ozonated olive oil as pulp capping material in non-vital primary molars.

Thus, the main purpose of this study is to evaluate and compare the clinical and radiographic effect of zinc oxide-ozonated olive oil versus Modified Triple Antibiotic Paste (MTAP) utilizing LSTR technique in the treatment of non-vital primary molars.

ELIGIBILITY:
Inclusion Criteria: 1- Cooperative patients in the age group of (4-7) years with no associated systemic illness.

2- Bilateral mandibular primary molars showing signs and symptoms of pulp necrosis or chronic pulp infection with/without hemorrhage, suppuration, or purulence.

3- Spontaneous pain or tenderness to percussion. 4- Presence of chronic apical abscess, sinus tract, or grade I mobility. 5-The tooth should be restorable. 6- Radiographic characteristics are:

1. Widening of Periodontal ligament space.
2. Radicular involvement.
3. Furcation involvement less than or equal to half of the shortest root in the vertical dimension

   -

   Exclusion Criteria: Exclusion criteria :
   1. Physiologic root resorption is more than one-third of its length.
   2. Excessive internal resorption.
   3. Non-restorable teeth exhibiting greater than grade I mobility.
   4. Perforation into the bifurcation.
   5. Any underlying pathological lesion.
   6. Any previous history of allergy to the antibiotics used in the study. -

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
primary out come | 3,6,9,12 months
  .evaluate clinical outcomes including Absence of pain or tenderness, No tooth mobility, and Presence of healthy soft tissue; no swelling, redness, or sinus tract for both groups including zinc oxide ozonated oil group and MTAP group during the follow-up periods 3,6,9,12 months follow up evaluate radiographic effect of both materials on: Continuity of lamina Dura, Static or reduction in the size of existing pathologic intra-radicular or periapical radiolucency., No newly formed radiographic lesion, Absence of pathological root resorption, and Evidence of bone regeneration utilizing gray value
primary outcome | 3,6,9,12 months follow up
  evaluate radiograhic effect of both materials on :
  * Continuity of lamina Dura.
  * Static or reduction in the size of existing pathologic intra-radicular or periapical radiolucency.
  * No newly formed radiographic lesion.
  * Absence of pathological root resorption
  * Evidence of bone regeneration utilizatig gray value

SECONDARY OUTCOMES:
secondary out come | 12 months follow up
  evaluate lesion sterlization and tissue repair by (Zn-OO)as a substitute to pulpectomy

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Sh El-Desokey, Professor, Principal Investigator — Faculty of dentistry Tanta university , tanta; Fatma el hendawy, Professor, Study Director — Faculty of dentistry Tanta university , Tanta; Nancy metwally, doctor, Study Director — Faculty of dentistry Tanta university , Tanta
Locations (2):
- Egypt (2):
  - Faculty of dentistry Tanta university, Tanta, Gharbia Governorate
  - Nouran Esmail Mohamed Shalaby, Menouf